CLINICAL TRIAL: NCT03852264
Title: Oxytocin Pathways and the Health Effects of Human-Animal Interaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1808883345
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-03

CONDITIONS: Human-Animal Bond; Human-Animal Interaction
Keywords: Oxytocin; Cortisol; Human-animal interaction
MeSH Terms: conditions — Human-Animal Bond; Human-Animal Interaction

STUDY DESIGN:
Intervention Model Description: Within-subjects, 3 conditions, 2 condition orders balanced across participants
Who Masked: Outcomes Assessor
Masking Description: Personnel analyzing hormones will be blinded to the experimental condition samples were collected from.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pet Dog Interaction first, then Nonsocial Control, then Unfamiliar Dog Interaction (Experimental): Participant's first study visit involved 25 minutes of interaction with the participant's pet dog. The second study visit involved 25 minutes of individual play with toys. The third study visit involved 25 minutes of interaction with an unfamiliar dog.
  Interventions: Behavioral: Pet dog; Behavioral: Unfamiliar dog; Behavioral: Nonsocial control
- Unfamiliar Dog Interaction first, then Nonsocial Control, then Pet Dog Interaction (Experimental): Participant's first study visit involved 25 minutes of interaction with an unfamiliar dog. The second study visit involved 25 minutes of individual play with toys. The third study visit involved 25 minutes of interaction with the participant's pet dog.
  Interventions: Behavioral: Pet dog; Behavioral: Unfamiliar dog; Behavioral: Nonsocial control

INTERVENTIONS:
Behavioral: Pet dog — Children will interact freely with their pet dog for 25 minutes.
Behavioral: Unfamiliar dog — Children will interact freely with an unfamiliar dog for 25 minutes
Behavioral: Nonsocial control — Children will play with age-appropriate toys/games for 25 minutes.

SUMMARY:
This study investigates the roles of oxytocin pathways in human-animal interaction.

DETAILED DESCRIPTION:
This study investigates the roles of oxytocin pathways in human-animal interaction. Children will participate in three conditions involving friendly interactions with dogs, or play with toys at a university laboratory. Child and dog saliva and urine will be assayed for oxytocin concentrations. We will assess variation in oxytocin concentrations in relation to different experimental conditions, and in relation to specific behaviors and psychological constructs.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study will include typically-developing children between 8-10 years who have lived with a companion dog in the household for at least 6 months.

Exclusion Criteria:

* known medical diseases or injuries involving the central nervous or endocrine systems, major physical abnormalities, seizures, and significant sensory, cognitive, or motor impairments, current use of psychoactive medications

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the local community through email listservs, print advertisements, social media, and flyers distributed to schools, libraries, museums, and veterinary clinics. Recruitment occurred between February 1, 2019 and February 1, 2022.
Pre-assignment Details: None / not applicable
Period: First Research Visit
Arm/Group | Pet Dog Interaction First, Then Nonsocial Control, Then Unfamiliar Dog Interaction | Unfamiliar Dog Interaction First, Then Nonsocial Control, Then Pet Dog Interaction
Started | 30 | 25
Completed | 30 | 25
Not Completed | 0 | 0
Period: Second Research Visit
Arm/Group | Pet Dog Interaction First, Then Nonsocial Control, Then Unfamiliar Dog Interaction | Unfamiliar Dog Interaction First, Then Nonsocial Control, Then Pet Dog Interaction
Started | 30 | 25
Completed | 30 | 25
Not Completed | 0 | 0
Period: Third Research Visit
Arm/Group | Pet Dog Interaction First, Then Nonsocial Control, Then Unfamiliar Dog Interaction | Unfamiliar Dog Interaction First, Then Nonsocial Control, Then Pet Dog Interaction
Started | 30 | 25
Completed | 29 | 25
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pet Dog Interaction First, Then Nonsocial Control, Then Unfamiliar Dog Interaction | Unfamiliar Dog Interaction First, Then Nonsocial Control, Then Pet Dog Interaction | Total
Number analyzed (Participants) | 30 | 25 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 25 | 55
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 18 | 13 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 3 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 22 | 27
Region of Enrollment [Number; unit: participants]
  United States | 30 | 25 | 55

OUTCOME MEASURES:

1. Primary Outcome: Salivary Oxytocin, Area Under the Curve
Description: Change from baseline measured as the area under the curve with respect to the initial value (AUCi).
Time Frame: baseline, 15 minutes
Population: All study participants for whom saliva samples were available for analysis
Measure: Mean (Standard Error); unit: pg/mL x minutes
Groups:
- Pet Dog Interaction: Participants interacted with their pet dog
- Unfamiliar Dog Interaction: Participants interacted with a dog who was unfamiliar to them
- Toys Interaction: Participants interacted with an assortment of toys
Arm/Group | Pet Dog Interaction | Unfamiliar Dog Interaction | Toys Interaction
Number analyzed (Participants) | 55 | 53 | 55
pg/mL x minutes | -3.03 (1.59) | -3.83 (1.67) | -5.57 (1.73)
Statistical Analysis 1: Comparison: Pet Dog Interaction vs Unfamiliar Dog Interaction vs Toys Interaction; Bayesian multilevel model of area under the curve with respect to initial value (AUCi) as a function of experimental condition; Test type: Other — 90% credible interval for contrast between conditions; Mean Difference (Net) = 2.61, 90% CI 2-sided [-1.29 to 6.38] — Contrast reflecting Pet Dog Interaction - Toys Interaction
Statistical Analysis 2: Comparison: Pet Dog Interaction vs Unfamiliar Dog Interaction vs Toys Interaction; [analysis description as in outcome 1, analysis 1]; Test type: Other — 90% credible interval for contrast between conditions; Mean Difference (Net) = 1.62, 90% CI 2-sided [-2.18 to 5.45] — Contrast reflecting Unfamiliar Dog Interaction - Toys Interaction
Statistical Analysis 3: Comparison: Pet Dog Interaction vs Unfamiliar Dog Interaction vs Toys Interaction; [analysis description as in outcome 1, analysis 1]; Test type: Other — 90% credible interval for contrast between conditions; Mean Difference (Net) = -1.00, 90% CI 2-sided [-4.93 to 2.83] — Contrast reflecting Unfamiliar Dog Interaction - Pet Dog Interaction

2. Primary Outcome: Urinary Oxytocin, Area Under the Curve
Description: Change from baseline measured as the area under the curve with respect to the initial value (AUCi).
Time Frame: baseline, 50 minutes
Population: All children with urine samples available for analysis
Measure: Mean (Standard Error); unit: pg/ml x minutes
Arm/Group | Pet Dog Interaction | Unfamiliar Dog Interaction | Toys Interaction
Number analyzed (Participants) | 52 | 46 | 50
pg/ml x minutes | 0.261 (0.372) | -0.219 (0.366) | -0.180 (0.407)
Statistical Analysis 1: Comparison: Pet Dog Interaction vs Unfamiliar Dog Interaction vs Toys Interaction; [analysis description as in outcome 1, analysis 1]; Test type: Other — 90% credible interval for contrast between conditions; Mean Difference (Net) = 0.3482, 90% CI 2-sided [-0.476 to 1.211] — Contrast reflecting Pet Dog Interaction - Toys Interaction
Statistical Analysis 2: Comparison: Pet Dog Interaction vs Unfamiliar Dog Interaction vs Toys Interaction; [analysis description as in outcome 1, analysis 1]; Test type: Other — 90% credible interval for contrast between conditions; Mean Difference (Net) = -0.0635, 90% CI 2-sided [-0.931 to 0.803] — Contrast reflecting Unfamiliar Dog Interaction - Toys Interaction
Statistical Analysis 3: Comparison: Pet Dog Interaction vs Unfamiliar Dog Interaction vs Toys Interaction; [analysis description as in outcome 1, analysis 1]; Test type: Other — 90% credible interval for contrast between conditions; Mean Difference (Net) = -0.4220, 90% CI 2-sided [-1.319 to 0.445] — Contrast reflecting Unfamiliar Dog Interaction - Pet Dog Interaction

3. Secondary Outcome: Salivary Cortisol, Area Under the Curve
Description: Change from baseline measured as the area under the curve with respect to the initial value (AUCi).
Time Frame: baseline, 50 minutes
Population: All participants with saliva samples available for analysis
Measure: Mean (Standard Error); unit: pg/mL x minutes
Arm/Group | Pet Dog Interaction | Unfamiliar Dog Interaction | Toys Interaction
Number analyzed (Participants) | 55 | 54 | 54
pg/mL x minutes | -99.7 (20.2) | -221.1 (70.1) | -103.0 (29.2)
Statistical Analysis 1: Comparison: Pet Dog Interaction vs Unfamiliar Dog Interaction vs Toys Interaction; [analysis description as in outcome 1, analysis 1]; Test type: Other — 90% credible interval for contrast between conditions; Mean Difference (Net) = 0.468, 90% CI 2-sided [-101 to 99.5] — Contrast reflecting Pet Dog Interaction - Toys Interaction
Statistical Analysis 2: Comparison: Pet Dog Interaction vs Unfamiliar Dog Interaction vs Toys Interaction; [analysis description as in outcome 1, analysis 1]; Test type: Other — 90% credible interval for contrast between conditions; Mean Difference (Net) = -115, 90% CI 2-sided [-225 to -15.5] — Contrast reflecting Unfamiliar Dog Interaction - Toys Interaction
Statistical Analysis 3: Comparison: Pet Dog Interaction vs Unfamiliar Dog Interaction vs Toys Interaction; [analysis description as in outcome 1, analysis 1]; Test type: Other — 90% credible interval for contrast between conditions; Mean Difference (Net) = -115.48, 90% CI 2-sided [-223 to -16.2] — Contrast reflecting Unfamiliar Dog Interaction - Pet Dog Interaction

4. Secondary Outcome: Urinary Vasopressin, Area Under the Curve
Description: Change from baseline measured as the area under the curve with respect to the initial value (AUCi).
Time Frame: baseline, 50 minutes
Population: unable to complete assay for this outcome
Arm/Group | Pet Dog Interaction | Unfamiliar Dog Interaction | Toys Interaction
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 hour
Groups:
- Pet Dog Interaction: Participants interacted with their pet dog for 25 minutes
- Unfamiliar Dog Interaction: Participants interacted with an unfamiliar dog for 25 minutes
- Toys Interaction: Participants interacted with an assortment of toys for 25 minutes
Arm/Group | Pet Dog Interaction | Unfamiliar Dog Interaction | Toys Interaction
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03852264/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT03852264/ICF_001.pdf